CLINICAL TRIAL: NCT02276742
Title: Lifestyle Management of CKD in Obese Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 14-01469; 14-A0-00-002990-01 (Other Grant/Funding Number: NIH/NIDDK)
Record Dates: First submitted 2014-09-12; First posted 2014-10-28 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Obesity; Type 2 Diabetes; Chronic Kidney Disease (CKD)
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual Care (UC) (No Intervention): Participants randomized to UC will receive baseline advice about the value of losing weight, becoming more physically active, and limiting intake of sodium and inorganic phosphates followed by 12 mos of UC. We have elected not to use a control group in which we provide equivalent attention to both study arms. Behaviors are difficult to change and there is no reason to believe that simply giving participants attention would create behavioral changes sufficient to result in weight loss, reduce sodium excretion, or reduce serum phosphorus. Numerous weight loss studies, including Look AHEAD, have used attention control groups that did not demonstrate weight loss.
- Social Cognitive Theory (SCT) (Active Comparator): Participants will be exposed to a group behavioral intervention that is based on SCT, which focuses on the role played by self-referent thought in the maintenance of behavior change. Self- efficacy is derived from four major sources of information: mastery experiences, social modeling, verbal persuasion, and physiological states. Mastery experiences will include emphasizing past successes; setting incremental, easily achievable goals; identifying modifiable barriers to healthy behavior; receiving positive feedback on goal achievement; and practicing problem solving skills around barriers to adherence.
  Interventions: Behavioral: Social Cognitive Theory
- Monitoring (Active Comparator): Participants will be taught how to use a lifestyle self-monitoring program to reduce information processing requirements, make readily available the information required to make good self-management decisions, deliver automated, real-time feedback about achievement of behavioral goals, and permit individualized guidance from an interventionist who uses the MyNetDiary® electronic log to provide targeted education and advice. The Monitoring intervention reduces information processing demands by making relevant nutritional information readily available. Technology-based self-monitoring also can be used by interventionists to reduce information processing burden by using it for targeted counseling
  Interventions: Other: Monitoring
- Combined (Active Comparator): Participants randomized to COMBINED will receive all aspects of the SCT and MONITORING intervention conditions. Social Cognitive Theory based behavioral intervention in complex patients is strengthened when technology is used to manage information complexity, and weakened in its absence. The Monitoring intervention reduces information processing demands by making relevant nutritional information readily available. Technology-based self-monitoring also can be used by interventionists to reduce information processing burden by using it for targeted counseling
  Interventions: Behavioral: Social Cognitive Theory; Other: Monitoring

INTERVENTIONS:
Behavioral: Social Cognitive Theory — focuses on the role played by self-referent thought in the maintenance of behavior change. Self- efficacy (e.g., the participant's confidence in their ability to engage in healthier behavior) is derived from four major sources of information: mastery experiences, social modeling, verbal persuasion, and physiological states
  Other Names: SCT
  Arms: Combined; Social Cognitive Theory (SCT)
Other: Monitoring — Technology-based self-monitoring reduces information processing demands by making relevant nutritional information readily available. Technology-based self-monitoring also can be used by interventionists to reduce information processing burden by using it for targeted counseling. For example, simultaneous consideration of all pertinent dietary recommendations would likely be overwhelming for an obese person with diabetes and CKD. By using an electronic log accessible to the interventionist, such a person could initially focus on calorie restrictions, with the interventionist stepping-in when problematic behaviors become evident.
  Other Names: Technology-based self-monitoring
  Arms: Combined; Monitoring

SUMMARY:
The purpose of this randomized clinical trial is to evaluate the efficacy of 3 different technology-supported approaches to engaging 300 individuals with diabetes and concurrent chronic kidney disease in weight loss, dietary sodium restriction, and dietary restriction of inorganic phosphates when compared to usual care. Participants will be randomized to 1 of 4 groups, Usual Care (UC), Social Cognitive Theory-based Group Counseling (SCT), Mobile self-monitoring with tailored feedback and counseling (MONITORING), or a combination of SCT plus MONITORING conditions (COMBINED). Investigators will evaluate the intervention arms primarily in terms of weight reduction, urinary sodium excretion, and serum phosphorus and, secondarily in terms of physical activity, blood pressure, fasting lipids, medication requirements, and pulse wave velocity. Measurements will occur at baseline, 6, and 12 months. The statistical modeling of the baseline, 6 mos and 12 mos outcome variables will be based on logistic generalized linear mixed models (for binary outcomes) linear mixed models (for continuous outcomes), and random effects multinomial models (for outcomes with more than 2 levels, such as changes in medication management). In separate analyses of the intervention arm only, investigators will model self-monitoring adherence and examine possible associations between self-monitoring adherence and outcomes. The mediating effect of self-efficacy on the primary outcomes will be evaluated using structural equation models.

DETAILED DESCRIPTION:
Investigators will conduct a 2x2 factorial, randomized clinical trial. All participants will receive usual care. Prior to randomization, participants will be stratified by recruitment siteParticipants will be randomized to 1 of 4 groups, Usual Care (UC), Social Cognitive Theory-based Group Counseling (SCT), Mobile self-monitoring with tailored feedback and counseling (MONITORING), or a combination of SCT plus MONITORING conditions (COMBINED). Investigators will evaluate the intervention arms primarily in terms of weight reduction, urinary sodium excretion, and serum phosphorus and, secondarily in terms of physical activity, blood pressure, fasting lipids, medication requirements, and pulse wave velocity. Measurements will occur at baseline, 6, and 12 months. The statistical modeling of the baseline, 6 mos and 12 mos outcome variables will be based on logistic generalized linear mixed models (for binary outcomes) linear mixed models (for continuous outcomes), and random effects multinomial models (for outcomes with more than 2 levels, such as changes in medication management). In separate analyses of the intervention arm only, investigators will model self-monitoring adherence and examine possible associations between self-monitoring adherence and outcomes. The mediating effect of self-efficacy on the primary outcomes will be evaluated using structural equation models

II. CHARACTERISTICS OF THE RESEARCH POPULATION

1. Number of subjects. Investigators will recruit 300 participants to the study. Investigators will focus our study on those with diabetic CKD as this form of the disease progresses more rapidly than other forms of CKD. Focusing on diabetic CKD also allows us to expand logically upon Look AHEAD, and build upon our work in T2DM patients with the ENHANCE study. Investigators will recruit participants from 3 clinical sites in New York City: Nephrology Family Group Practice at NYU Langone Medical Center (NYULMC), the Bellevue Hospital Diabetes Clinic, and New York Harbor VA. Preliminary data from these 3 practice settings indicate that investigators will have access to 4,292 potentially eligible patients from which investigators must recruit only 7.0% to enroll 300. Our prior studies suggest that investigators will retain 80% resulting in a final sample of 240. Investigators are projecting 64 participant measurement visits in Year 1; 248 in Year 2; 288 in Year 3; 244 in Year 4; and 56 in Year 5.

Unless otherwise noted, measurements occur at baseline, 6, and 12 mos. Data are collected with visits to NYU Clinical and Translational Resource Center (CTRC). Information to be obtained from participants at each visit includes height and weight, serum and urine samples; blood pressure; investigator administered instruments (sociodemographics, comorbid conditions, Mini Mental Status Exam, and self-efficacy instruments), medication inventories, and Pulse Wave Velocity. Eight blood tests will be performed: cystatin-C, lipids, phosphorus, calcium, PTH or parathyroid hormone, vitamin D, pre-albumin and albumin. These tests are estimated to require, in total, approximately 45 mls (of blood.

One week before their scheduled measurement visit, a 24-hour urine specimen container and instructions for collection are mailed to the participant. Participants are contacted 2 days prior to their appointment to remind them of their measurement visit, collect their urine, fast, and abstain from caffeine for 12 hours prior to their appointment. Laboratory tests are collected, spun, refrigerated, batched and sent for processing in the CLIA-certified NYU CTSI Translational Research Laboratories by personnel blinded to group assignment. The PWV of the brachial-ankle (baPWV) and carotid-femoral (cfPWV) will be collected by trained research associates at the CTRC.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible for the study, the individual must be 40 years of age or older
* Have a DRG Code of T2DM, GFR of 15-89 ml/min/1.73m2 and a BMI >30 kg/m2.
* The participant's physician of record will have verified that his/her patient can safely participant in an intervention study that involves weight loss and a goal of 150 minutes/week of moderate physical activity comparable to brisk walking.

Exclusion Criteria:

* Investigators will exclude from participation those with the following characteristics:

  1. unable or unwilling to provide informed consent
  2. unable to participate meaningfully in an intervention that involves group sessions (e.g., due to uncorrected hearing impairment, non-English-speaking)
  3. unable to read or otherwise use an iPad to monitor dietary intake, physical activity, and weight (e.g., blind, illiterate)
  4. unwilling to accept randomization assignment
  5. pregnant, or plans to become pregnant in the next 12 months, less than 3 months postpartum, or nursing or within 6 weeks of having completed nursing
  6. weight loss of > 10% in the past 6 months except for postpartum weight loss
  7. unable to walk 0.25 miles in 10 minutes
  8. a major psychiatric disorder
  9. planning gastric bypass surgery in the next 12 months
  10. individuals who are institutionalized (e.g., in a nursing home or personal care facility, or those who are incarcerated and have no control over their diet).
* Investigators will exclude from the study those with underlying diseases that would increase the risk of participating in an intervention involving caloric restriction and physical activity.
* Such individuals would include those requiring treatment for cancer, exclusive of skin cancer other than melanoma, in the past 2 years; infectious diseases including untreated AIDS and active tuberculosis; uncontrolled hypertension of >190 mmHg SBP or >105 mmHg DBP despite treatment; stroke or TIA in the past 6 months; conditions requiring the use of home oxygen; or other chronic disease or condition likely to limit life span to < 1 year.
* Because of the dietary requirements of a pregnant woman, and the nature of weight loss and gain with pregnancy, inclusion of pregnant women in the study would confound the study results. Those who become pregnant during the study will be withdrawn from the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
Weight in kgs will be obtained using a single, calibrated scale | Change from baseline in weight at 6 months
  Compared to the UC group, SCT and COMBINED groups will demonstrate a greater proportion of participants losing at least 5% of their baseline weight at 6 months, with these differences sustained at 12 months.
Serum phosphorus will be evaluated from a venipuncture sample | Change from baseline in Serum Phosphourous at 6 months
  Compared to the UC group, SCT and COMBINED groups will demonstrate larger reductions in serum phosphorus, with reductions sustained at 12 months.
Urinary sodium will be determined from a time 24-hour urine sample | Change from baseline in Urinary sodium at 6 months
  Compared to the UC group, SCT and COMBINED groups will demonstrate larger reductions in urinary sodium excretion, with reductions sustained at 12 months
Weight in kgs will be obtained using a single, calibrated scale | Change from baseline in weight at 12 months
Serum phosphorus will be evaluated from a venipuncture sample | Change from baseline in Serum phosphorus at 12 months
Urinary sodium will be determined from a time 24-hour urine sample | Change from baseline in Urinary sodium at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann Sevick, ScD, RN, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Cashmore BA, Cooper TE, Evangelidis NM, Green SC, Lopez-Vargas P, Tunnicliffe DJ. Education programmes for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 Aug 22;8(8):CD007374. doi: 10.1002/14651858.CD007374.pub3. PMID 39171639
- [Derived] McMahon EJ, Campbell KL, Bauer JD, Mudge DW, Kelly JT. Altered dietary salt intake for people with chronic kidney disease. Cochrane Database Syst Rev. 2021 Jun 24;6(6):CD010070. doi: 10.1002/14651858.CD010070.pub3. PMID 34164803
- [Derived] Conley MM, McFarlane CM, Johnson DW, Kelly JT, Campbell KL, MacLaughlin HL. Interventions for weight loss in people with chronic kidney disease who are overweight or obese. Cochrane Database Syst Rev. 2021 Mar 30;3(3):CD013119. doi: 10.1002/14651858.CD013119.pub2. PMID 33782940
- [Derived] Sevick MA, Woolf K, Mattoo A, Katz SD, Li H, St-Jules DE, Jagannathan R, Hu L, Pompeii ML, Ganguzza L, Li Z, Sierra A, Williams SK, Goldfarb DS. The Healthy Hearts and Kidneys (HHK) study: Design of a 2x2 RCT of technology-supported self-monitoring and social cognitive theory-based counseling to engage overweight people with diabetes and chronic kidney disease in multiple lifestyle changes. Contemp Clin Trials. 2018 Jan;64:265-273. doi: 10.1016/j.cct.2017.08.020. Epub 2017 Sep 1. PMID 28867396